CLINICAL TRIAL: NCT02652377
Title: A Randomized, Double-Blind, Pbo-Controlled, Study of EDP-494 to Evaluate the Safety and PK of SAD/FE in Healthy Subjects and MAD in Healthy and in Subjects With CHC Infection (POC)
Brief Title: EDP-494-001: A Study of EDP-494 in Healthy Subjects and Hepatitis C Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP-494-001
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- EDP-494 SAD Cohorts (Experimental): EDP-494, oral 50 mg, 100mg, 200mg, 400mg and 800 mg, capsules, once daily in one single administration
  Interventions: Drug: EDP-494
- EDP-494 MAD/POC Cohorts (Experimental): EDP-494, oral 200mg, 400mg and 800 mg, capsules, once daily for 14 days
  Interventions: Drug: EDP-494
- EDP-494 SAD Placebo Cohort (Placebo Comparator)
  Interventions: Drug: Placebo
- EDP-494 MAD/POC Placebo Cohort (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-494 — 10, 100 and 200 mg capsules
  Arms: EDP-494 MAD/POC Cohorts; EDP-494 SAD Cohorts
Drug: Placebo — placebo to match EDP-494
  Arms: EDP-494 MAD/POC Placebo Cohort; EDP-494 SAD Placebo Cohort

SUMMARY:
This randomized, double-blind study will assess the safety, pharmacokinetics and efficacy of a single and multiple dose(s) of orally QD administered EDP-494 in healthy volunteers (HV) and in treatment-naive subjects with GT1/3 chronic hepatitis C (CHC) infection.

DETAILED DESCRIPTION:
The first phase explores single ascending doses of EDP-494 (active drug or placebo) in healthy subjects. A 'fasted' vs 'fed' two-part cohort will also assess food effect.

The second phase involves multiple ascending doses (active drug or placebo) for 14 days in healthy subjects.

The third, proof of concept, phase will assess two different doses for 14 days each in Hepatitis C patients.

Each cohort within each phase will consist of 8 subjects randomized to either EDP-494 or placebo in a 3 to 1 ratio, with the exception of the food effect cohort, which will consist of 10 subjects randomised in a 4 to 1 ratio.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers (SAD and MAD Phases):

* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Female subjects must be of non-childbearing potential.
* All male participants who have not had a vasectomy must use effective contraception from Day -1 to 90 days after their last dose of study drug.
* Body mass index of 18 to 30 kg/m2 with a minimum body weight of 50 kg.
* An informed consent document signed and dated by the subject.

Exclusion Criteria for Healthy Volunteers (SAD and MAD Phases):

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* History of regular alcohol consumption
* Participation in a clinical trial within 30 days prior to study drug administration.
* Use of prescription drugs, non-prescription drugs, dietary supplements, herbal supplements, hormonal therapy/replacement or CYP3A4 substrates, inducers and inhibitors within 14 days prior to the first dose of study medication

Inclusion Criteria for HCV-Infected Subjects (POC Phase):

* Males and females aged 18 years and less than 70 years.
* Female subjects must be of non-childbearing potential.
* All male participants who have not had a vasectomy must use effective contraception from Day -1 to 90 days after their last dose of study drug.
* Body mass index of 18 to 36 kg/m2 with a minimum body weight of 50 kg.
* Treatment naïve subjects with chronic HCV infection,
* HCV GT1 (including 1a, 1b, or mixed subtypes of GT1) or GT3.
* HCV RNA ≥100,000 IU/mL at screening.
* An informed consent document signed and dated by the subject.

Exclusion Criteria for HCV-Infected Subjects (POC Phase):

* Women of childbearing potential (WOCBP).
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug.
* A positive urine drug screen at screening unless on an approved prescription.
* History of participation in a clinical trial with a polymerase inhibitor or previous treatment with a polymerase inhibitor, where at least one dose of the polymerase inhibitor was consumed. Subjects who were dosed with placebo on a clinical trial may be enrolled in this study.
* Clinically significant electrocardiogram abnormalities or QTcF greater than 450 msec for males and 470 msec for females at either screening or baseline, or any prior history of QT abnormality.
* Co-infection with HIV-1, HIV-2 or HBV.
* Have clinically significant laboratory abnormalities at screening:

  * Absolute neutrophil count (ANC) < 1500/mm2 (1.5 x 109L)
  * Platelets <90,000/mm2 (90 x 109L)
  * Hemoglobin < 13g/dL for males and < 12g/dL for females
  * Serum creatinine >1.5 x upper limit of normal (ULN) or creatinine clearance < 50 mL/min; estimated by the cockcroft -Gault formula [(140-age) x weight (kg)/72 x serum creatinine (mg/dL), if female multiply by 0.85]
  * Total bilirubin greater than the ULN
  * Serum alanine transaminase (ALT) > 5 x ULN
  * Serum aspartate aminotransferase (AST) > 5 x ULN
  * Alkaline phosphatase > 1.25 x ULN
  * Pancreatic Amylase > 1.1 x ULN
  * Alpha fetoprotein (AFP) > 50 ng/mL unless a liver imaging study (CT, MRI) shows no clinically significant lesions within 6 months prior to the first dose of study drug.
* Patients with evidence of cirrhosis; cirrhosis is defined as any one of the following: a) any biopsy showing cirrhosis (Knodell score <3, Metavir score <3, Ishak score <4); b) Fibroscan evaluation within 6 months prior to screening with a liver stiffness score of ><12.5 kPa.
* Other significant, unstable or uncontrolled medical history, such as neurological, endocrine, malignancy, renal, psychiatric, respiratory, cardiac, gastrointestinal, allergic, immunological, etc. disease.
* Use of concomitant medications, including vitamins or herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
Composite number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG, and abnormal clinical laboratory results administered to healthy volunteers and multiple doses of EDP-494 | From screening and baseline to the 4 week follow-up visit
  Tabulation of the number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG, echo and abnormal clinical laboratory results (including chemistry, hematology, and urine).
  Administered to healthy volunteers and multiple doses of EDP-494 administered to healthy volunteers and subjects with Chronic Hepatitis C (CHC) genotype 1 and 3 infection

SECONDARY OUTCOMES:
Cmax | 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, 72 (Day 4), 96 (Day 5), 120 (Day 6)*, 144 (Day 7) and 168 (Day 8) hrs postdose
  EDP-494 and metabolites
Cmax | Day 1: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15 hrs; Days 2, 3, 5, 7, 9, 12: 0 (Predose); Day 14: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, 72, 96, 120, 144 and 168 hrs postdose
  EDP-494 and metabolites
AUC | 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, 72, 96, 120*, 144, and 168 hrs postdose
  EDP-494 and metabolites
AUC | Day 1: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15 hrs; Days 2, 3, 5, 7, 9, 12: 0 (Predose);Day 14: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, 72, 96, 120, 144 and 168 hrs postdose
  EDP-494 and metabolites
Change from baseline in plasma HCV RNA (log10 IU/mL) | Baseline up to 14 days
Amino Acid Changes in HCV polymerase NS5b | Baseline up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Gane, MD, Principal Investigator — Auckland Clinical Studies (ACS),
Locations (1):
- Auckland Clinical Studies Ltd, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
Once the clinical study report has been submitted to the appropriate Regulatory authorities, a lay person summary will be provided to all study subjects by mail or email.